CLINICAL TRIAL: NCT03916133
Title: Evaluation of the Clinical Feasibility of Angiographic Flat-detector CT (FDCT) Perfusion Imaging (6sPBV) Technique.
Brief Title: Analysis of Selective Cerebrovascular Distribution With FDCT in the Angiosuite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Thijs van der Zijden, Principal Investigator, University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18/17/222
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Ischemic Stroke; Intracranial Aneurysm; Intracranial Arterial Diseases; Cerebral Hypoxia; Intracranial Vascular Disorder
MeSH Terms: conditions — Ischemic Stroke; Intracranial Aneurysm; Intracranial Arterial Diseases; Hypoxia, Brain; Cerebrovascular Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Other): Included patients will undergo angiographic FDCT perfusion imaging.The study will be embedded in the standard procedure of pre-operative diagnostics and angiographic control after EC-IC bypass treatment of steno-occlusive disease and during pre-embolization mapping and embolization procedure. An informed consent will be acquired during consultations in the preparatory process of the different examinations and treatments
  Interventions: Diagnostic Test: Intervention group

INTERVENTIONS:
Diagnostic Test: Intervention group — 6s PBV mapping will be conducted
  Other Names: Flat-detector CT perfusion imaging

SUMMARY:
The aim of this study is to evaluate the clinical feasibility of the angiographic Flat Detector CT perfusion imaging (6s PBV) technique. The investigators will examine the specific vessel distribution of patients with steno-occlusive disease, treated with a surgical extracranial-intracranial bypass and assess the cerebral perfusion during test occlusion upon a neurovascular treatment and in intracranial tumor patients referred for potential pre-operative embolization.

This study encompasses three scientific objectives:

1. What is the selective contribution of an individual bypass artery to the brain perfusion?
2. Is a selective intra-arterial angiographic perfusion examination useful in the decision-making of performing pre-operative embolization of intracranial tumors?
3. What is the usefulness of performing additive 6s PBV images compared to classical 2D angiography and/or clinical neurological evaluation in case of test occlusion in the evaluation of possible mother vessel occlusion in treatment of complex neurovascular diseases?

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for diagnostics and surgical (extracranial-intracranial bypass) treatment of steno-occlusive neurovascular disorders.
* Patients referred for hypervascular intracranial tumor resection
* Patients referred for angiographic test occlusion as part of treatment of complex neurovascular disorders.

Exclusion Criteria:

* Pregnant women or women trying to get pregnant
* People younger than 18 years old
* Patients with thyroid disorders and diabetes, especially those using medication with metformin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Performance of flat-detector CT imaging in angiosuite | 1 day
  The quality of the imaging scans obtained with FDCT will be assessed compared to conventional imaging techniques (CT, angiography and MRI)

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Antwerp, België, Belgium

IPD SHARING:
Plan to Share IPD: No